CLINICAL TRIAL: NCT01452022
Title: A Prospective Open-label Non-randomdised Multi-centre Clinical Study to Evaluate the Performance of Inductigraft in Posterolateral Fusion
Brief Title: Performance of Inductigraft in Spinal Fusion
Acronym: APOLLO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: Apatech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INDOUS1001
Record Dates: First submitted 2011-10-05; First posted 2011-10-14 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Degenerative Disk Disease; Spinal Stenosis of Lumbar Region
Keywords: inductigraft; osteoinductive; synthetic bone graft; posterolateral lumbar fusion; post market; lumbar spinal stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inductigraft (Experimental): open label non randomised to assess performance of synthetic bone graft using the product, Inductigraft, in posterolateral lumbar fusion
  Interventions: Device: Inductigraft

INTERVENTIONS:
Device: Inductigraft — Synthetic bone graft

SUMMARY:
This is an open-label non-randomised, prospective, post market study to evaluate the performance of Inductigraft (osteoinductive synthetic bone graft) in patients receiving posterolateral lumbar spine fusion through assessment of successful fusion at 12 months post operation using x-rays and CT scans. Quality of life questionnaires also used to assess clinical outcome measures such as pain and quality of life. Patients followed up for 24 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Degenerative Disk Disease (DDD) or lumbar spinal stenosis at one or two continuous spinal level(s), including subjects with spondylolisthesis (i.e. degenerative or isthmic)
* Has failed at least six months of non-operative treatment prior to clinical trial enrolment and is a candidate for spinal fusion surgery over one or two vertebral levels between, and including, L2 to S1 (i.e. second lumbar to first sacral)
* ≥ 18 years old and skeletally mature (epiphyses closed)
* Is, in the Investigator's opinion, psychosocially, mentally, and physically able to fully comply with this protocol, including the post-operative regimen, required follow up visits, the filling out of required forms, and have the ability to understand and give written informed consent.

Exclusion Criteria:

* Has diagnosis of symptomatic DDD, spondylolisthesis, or lumbar spinal stenosis at more than two levels
* Has had prior fusion surgery at any lumbar level
* Has systemic infection or infection at the surgical site
* History of significant metabolic bone disease such as osteomalacia, autoimmune disease including rheumatoid arthritis, renal disease, hepatic disease, peripheral vascular disease, insulin dependent diabetes, Paget's disease at the involved spinal level(s) or upper motor neuron disease (positive Babinski sign)
* Has a medical condition that would interfere with post-operative assessments and care (i.e. psychiatric disease, paraplegia, quadriplegia, etc.)
* Is in poor general health or any concurrent disease process that would place the subject in excessive risk to surgery (e.g. significant circulatory, pulmonary problems, or cardiac disease)
* Has a history (present or past) of substance abuse (recreational drugs, prescription drugs or alcohol) that in the Investigator's opinion may interfere with protocol assessments and/or with the subject's ability to complete the protocol required follow up
* Is known to be pregnant/breastfeeding at the time of enrollment, or plans to become pregnant during the course of the clinical trial
* Is participating in, or has completed within the last 30 days, another investigational clinical trial, which could confound results
* Has had three or more prior decompressive surgeries, or a prior posterior lumbar surgery resulting in significant muscle/ligament morbidity. This does NOT include facet saving techniques such as discectomy, laminotomy, and intradiscal procedures including nucleotomy, IDET procedures or annuloplasty procedures
* Has back or leg pain of unknown cause
* Morbid obesity defined as a Body Mass Index (BMI) ≥ 40
* Non-discogenic or non-stenotic cause of symptoms (e.g. tumour or fracture at the involved level)
* Has a condition or requires post-operative medications that may interfere with bone/soft tissue healing (i.e. oral or parenteral glucocorticoids, immunosuppressives, methotrexate, etc.), or that effect the rate of bone metabolism unless they have undergone a 14 day wash out period prior to surgery
* Is undergoing treatment for osteoporosis (excluding osteopenia) such that in the Investigator's opinion, spinal instrumentation would be contraindicated
* Is involved in on-going litigation, concerning their medical condition.
* Has a known allergy to silicon.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2011-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Fusion rate | 12 months after surgery
  Assessed by x-ray and CT scan

SECONDARY OUTCOMES:
Fusion rate | 6 and 24 months after surgery
  fusion rate at 6 and 24 months by x-ray/CT scan
Clinical Outcome Measure - pain | 6, 12 and 24 months
  Assessed by VAS scores
Clinical Outcome measure - Quality of Life | 6,12,and 24 months
  Oswestry Disability Index
Clinical Outcome measure - Quality of Life | 6,12,and 24 months
  SF-36 v2 short form, health questionnaire
Adverse events | 0-24 months after surgery
  Assessment of Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ciaran Bolger, Principal Investigator — Beaumont Hospital, Dublin
Locations (15):
- Germany (3):
  - Universitätsklinikum Bonn, Bonn
  - University of Cologne, Cologne
  - Ludwig-Maximilians-Universität München, München
- Hungary (2):
  - Buda Health Center, Budapest
  - University of Debrecen, Debrecen
- Beaumont Hospital, Dublin, Dublin, Ireland
- Spain (3):
  - Fundacio Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinical de Barcelona & Clinical Corachan, Barcelona
  - HGU Gregorio Marañón, Madrid
- United Kingdom (6):
  - University Hospital of Wales, Cardiff
  - Queens Medical Centre, Nottingham
  - Royal Preston Hospital, Preston
  - Salford Royal NHS Foundation Trust, Salford
  - Shire Southhampton Hospital, Southhampton
  - Musgrove Park Hospital, Tauton

REFERENCES:
- [Derived] Bolger C, Jones D, Czop S. Evaluation of an increased strut porosity silicate-substituted calcium phosphate, SiCaP EP, as a synthetic bone graft substitute in spinal fusion surgery: a prospective, open-label study. Eur Spine J. 2019 Jul;28(7):1733-1742. doi: 10.1007/s00586-019-05926-1. Epub 2019 Mar 5. PMID 30834972